CLINICAL TRIAL: NCT03650153
Title: Randomized Controlled Trial of MRI Target Biopsy: Transrectal vs. Transperineal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Al-Johara Al-Ibrahim Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Danny Rabah Study 2018
Record Dates: First submitted 2018-08-27; First posted 2018-08-28 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trans-rectal MRI targeted Biopsy (Active Comparator): Trans-rectal to perform the prostate MRI targeted biopsy The puncture points are at the rectal
  Interventions: Procedure: Trans-rectal MRI targeted Biopsy
- Trans-perineal MRI targeted Biopsy (Active Comparator): Trans-perineal to perform the prostate MRI targeted biopsy The puncture points are at the perineal
  Interventions: Procedure: Trans-perineal MRI targeted Biopsy

INTERVENTIONS:
Procedure: Trans-rectal MRI targeted Biopsy — Trans-rectal biopsy of the prostate: A procedure in which a sample of tissue is removed from the prostate using a thin needle that is inserted through the rectum and into the prostate.
  Arms: Trans-rectal MRI targeted Biopsy
Procedure: Trans-perineal MRI targeted Biopsy — Trans-perineal biopsy of the prostate: The sample is removed with a thin needle that is inserted through the skin of the perineum and into the prostate.
  Arms: Trans-perineal MRI targeted Biopsy

SUMMARY:
This prospective study of comparing between Transrectal and transperineal prostate MRI targeted biopsy to provide evidence for clinicians to select the appropriate biopsy approach under different conditions.

DETAILED DESCRIPTION:
This prospective study of comparing transperineal (TP) prostate MRI targeted biopsy with transrectal (TR) prostate MRI targeted biopsy was aimed to provide evidence for clinicians to select the appropriate biopsy approach under different conditions. TP (n = 75) and TR (n = 75) will be performed randomly for 150 patients who are suspicious of prostate cancer (PCa). The cancer detection rate (CDR), complication rate, visual analog scale (VAS) score, most painful procedure, number of repeated biopsy and additional anesthesia, and operating time (starting from lying down on the operating table to getting up) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* prostate-specific antigen > 4ng/ml
* Palpation is positive

Exclusion Criteria:

* older than 80y
* prostate-specific antigen > 100 ng/ml

Max Age: 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
the rate of positive detections | 1 year
  the rate of positive detections (How many case are Prostate cancer positive)

SECONDARY OUTCOMES:
the incidence rate of each complication | 1 year
  the Incidence of complication rate is the number of complications divided by the number of patients and the number of patients with complications. Complications were separated into those with major or minor sequelae and the proportion of each type that were due to medical error (avoidable).

OTHER OUTCOMES:
Pain level assessed by visual analogue scale (VAS) | 1 year
  The pain VAS is a unidimensional measure of pain intensity used adult populations.
  The pain VAS is a continuous scale comprised of a horizontal (HVAS) or vertical (VVAS) line, usually 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme. Instructions, time period for reporting, and verbal descriptor anchors have varied widely in the literature depending on intended use of the scale.
  Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100.
  A higher score indicates greater pain intensity. Based on the distribution of pain VAS scores in postsurgical patients who described their postoperative pain intensity as none, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75- 100 mm).

CONTACTS AND LOCATIONS:
Overall Officials: danny M Rabah, FRCS, Principal Investigator — Surgery Department and Cancer Research Chair, College of Medicine, King Saud University, Saudi Arabia
Locations (1):
- King Khalid University Hospital, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided